CLINICAL TRIAL: NCT06568640
Title: Evaluation and Exploration of the Safety and Efficacy of Superselective Adrenal Arterial Embolization in Patients With Essential Refractory Hypertension: A Proof-of-Concept Study
Brief Title: Superselective Adrenal Arterial Embolization for Refractory Hypertension: A Proof-of-Concept Study
Acronym: SAAE-RH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifei Dong, Deputy Director of the Department of Cardiology, Second Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-109
Record Dates: First submitted 2024-08-18; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Superselective adrenal arterial embolization; Interventional therapy
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: The study design is a single-center, open-label, self-controlled, single-arm, prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional treatment group (Experimental): superselective adrenal arterial embolization
  Interventions: Procedure: Superselective adrenal arterial embolization

INTERVENTIONS:
Procedure: Superselective adrenal arterial embolization — Superselective adrenal arterial embolization is an operation to inject embolic agent into adrenal artery through catheter to embolize part of adrenal gland, so as to reduce the secretion of adrenal hormone and reduce blood pressure.
  Other Names: Adrenal artery ablation; catheter-based adrenal ablation; Transcatheter Arterial Ablation; Transarterial embolization; percutaneous adrenal arterial embolization; selective adrenal artery embolization

SUMMARY:
The subjects of this study were patients with essential refractory hypertension. The purpose of this study is to evaluate the safety and efficacy of superselective adrenal arterial embolization (SAAE) in patients with primary refractory hypertension and to explore the possibility of SAAE in patients with primary refractory hypertension.After the subject completes the SAAE, an 8-week follow-up will be conducted to assess the safety and effectiveness of the SAAE.

DETAILED DESCRIPTION:
The subjects of this study were patients with essential refractory hypertension. The study design was a single-center, open-label, self-controlled, single-arm, prospective study. The purpose of this study is to evaluate the safety and efficacy of superselective adrenal arterial embolization (SAAE) in patients with primary refractory hypertension and to explore the possibility of SAAE in patients with primary refractory hypertension.After the subject completes the SAAE, an 8-week follow-up will be conducted to assess the safety and effectiveness of the SAAE.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, no gender restrictions;
* Primary refractory hypertension: Taking three antihypertensive drugs, including a - diuretic, with an average office systolic blood pressure ≥150 mmHg measured three times;
* Duration of hypertension greater than 6 months;
* Standing plasma aldosterone and renin activity not below the lower limit of the unit's reference range;
* Signed informed consent form.

Exclusion Criteria:

* Morning cortisol level < 4.3 µg/dL; estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m²; serum potassium level > 5.5 mmol/L;
* Type 1 diabetes, uncontrolled hyperthyroidism, malignant arrhythmias, malignant tumors, decompensated heart failure, severe liver dysfunction, severe hematological diseases, severe obstructive sleep apnea syndrome, history of myocardial infarction, syncope, cerebral hemorrhage, or cerebral infarction within the past 3 months;
* Pregnant women or those planning to conceive within the next year;
* Presence of other severe organic diseases that would make the patient unable to tolerate superselective adrenal arterial embolization;
* Adrenal mass with a diameter exceeding 2 cm;
* Severe allergy to contrast agents;
* Patients enrolled or planning to participate in other clinical studies that could impact the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
24-hour mean systolic blood pressure | 8 weeks after SAAE
  ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Proportion of patients with non-refractory hypertension | 8 weeks after SAAE
  Describe how many patients are converted from refractory hypertension to non-refractory hypertension
24-hour mean diastolic blood pressure | 8 weeks after SAAE
  ambulatory blood pressure monitoring
Safety monitoring:Procedure-related complications | up to 8 weeks
  Procedure-related complications include but are not limited to the following: transient arrhythmia during the SAAE procedure, incidence of hypertensive encephalopathy; post-procedure complications such as pleural effusion, brachial artery pseudoaneurysm, brachial artery thrombosis, pancreatitis, and contrast-induced nephropathy.
Safety monitoring:Adrenal-related hormones | 8 weeks after SAAE
  Plasma aldosterone concentration, plasma renin activity, plasma cortisol concentration, corticotropin-releasing hormone level, blood catecholamine levels, sex hormone levels.
Safety monitoring:Kidney function | 8 weeks after SAAE
  Estimated Glomerular Filtration Rate
Safety monitoring:Plasma electrolyte levels | 8 weeks after SAAE
  Plasma potassium

OTHER OUTCOMES:
Daytime average systolic blood pressure | 8 weeks after SAAE
  Daytime average systolic blood pressure
Daytime average diastolic blood pressure | 8 weeks after SAAE
  Daytime average diastolic blood pressure
Nighttime average systolic blood pressure | 8 weeks after SAAE
  Nighttime average systolic blood pressure
Nighttime average diastolic blood pressure | 8 weeks after SAAE
  Nighttime average diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Yifei Dong, Doctor, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, China

IPD SHARING:
Plan to Share IPD: No